CLINICAL TRIAL: NCT04209101
Title: Medical Students and Psychoactive Substances Use: For Whom to Worry?
Brief Title: Medical Students and Psychoactive Substances Use
Acronym: NC
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0615
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Psychoactive Substances Consumption
Keywords: Medical student; Psychoactive substances; Alcohol; Tobacco; At risk consumption

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Medical students are heavy users of psychoactive substances, and even if levels of use vary depending on the universities, the average levels are higher than most other students.

In France, however, the use of licit or illicit substance has not been precisely described in medical students. The aim of this study was therefore to define the different modes of consumption of medical students.

Methods: This study was a cross-sectional survey in medical students from the University of Montpellier, and the investigators performed a cluster analysis of data. Both medical students and residents were included. Socio-demographic, medico-psychological and addictological data were collected.

ELIGIBILITY:
Inclusion criteria:

* students had to be aged 18
* to be medical students

Exclusion criteria:

- refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To be included, students had to be aged 18 or more and to be medical students
Sampling Method: Non-Probability Sample
Enrollment: 942 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Define the different modes of consumption | 1 day
  The aim of this study was therefore to define the different modes of consumption of medical students.

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Donnadieu-Rigole, MD PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC